CLINICAL TRIAL: NCT05934526
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Inhalation of Seralutinib for the Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: Efficacy and Safety of Seralutinib in Adult Subjects With PAH (PROSERA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GB002, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB002-3101; 2023-503614-80-00 (Other: EU-CT number)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: seralutinib; GB002; PROSERA
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo inhaled orally twice daily (BID) up to 48 weeks
  Interventions: Drug: Placebo; Device: Generic Dry Powder Inhaler
- Seralutinib 90 mg (Experimental): Seralutinib inhaled orally BID up to 48 weeks
  Interventions: Drug: Seralutinib; Device: Generic Dry Powder Inhaler

INTERVENTIONS:
Drug: Placebo — Matching capsule containing placebo
  Arms: Placebo
Drug: Seralutinib — Capsule containing seralutinib
  Arms: Seralutinib 90 mg
Device: Generic Dry Powder Inhaler — Generic dry powder inhaler for seralutinib or placebo delivery

SUMMARY:
The primary objective of the study is to determine the effect of seralutinib on improving exercise capacity in subjects with WHO Group 1 PAH who are FC II or III. The secondary objective for this trial is to determine time to clinical worsening.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18 to 75 years.
2. Body mass index (BMI) ≥ 15 kg/m^2 and ≤ 40 kg/m^2.
3. Diagnosis of PAH classified by one of the following:

   1. Idiopathic PAH (IPAH) or heritable PAH (HPAH).
   2. PAH associated with connective tissue disease (CTD-APAH); PAH associated with anorexigen or PAH associated with methamphetamine use.
   3. Congenital heart disease with simple systemic to pulmonary shunt at least 1 year after surgical repair.
4. 6MWDs ≥ 150 meters and ≤ 475 meters during Screening prior to randomization.
5. WHO FC II or III.
6. US Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) Lite 2 Risk Score ≥ 5 OR NT-proBNP ≥ 300 ng/L OR PVR ≥ 800 dyne s/cm^5.
7. Cardiac catheterization within the screening period, or a standard of care right heart catheterization (RHC) (with pressure wave forms available for review) up to 48 weeks prior to Screening.

   1. Mean pulmonary arterial pressure (mPAP) > 20 mmHg (at rest), AND
   2. Pulmonary vascular resistance (PVR) ≥ 400 dyne·s/cm^5, AND
   3. Pulmonary capillary wedge pressure (PCWP) or left ventricle end-diastolic pressure (LVEDP) ≤ 15 mmHg.
8. Treatment with at least one allowed background PAH disease-specific medication prior to Screening.

   1. Subjects receiving treatment with endothelin receptor antagonists, phosphodiesterase type 5 inhibitors, guanylate cyclase stimulators, and/or prostacyclin analogues or prostacyclin receptor agonists are eligible only if on a stable dose for at least 12 weeks prior to and throughout Screening.
   2. Subjects receiving treatment with sotatercept are eligible only if on a stable dose of sotatercept for at least 24 weeks prior to and throughout Screening, with a RHC performed during Screening (or within 2 weeks prior to Screening).
9. Pulmonary function tests (PFTs) at Screening or completed no more than 12 weeks prior to Screening.
10. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and on Day 1 before first administration of Investigational Product (IP).
11. WOCBP who are not abstinent and intend to be sexually active with a non-sterilized male partner must be willing to use a highly effective method of contraception from consent through 30 days following the last administration of IP.
12. Male subjects: Non-sterilized male subjects who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom from consent through 90 days after the last dose of IP.

Exclusion Criteria:

1. Evidence of chronic thromboembolic disease or acute pulmonary embolism.
2. Uncontrolled systemic hypertension as evidenced by systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg.
3. Systolic blood pressure < 90 mm Hg during Screening.
4. WHO Pulmonary Hypertension Group 2 - 5.
5. Human immunodeficiency virus (HIV)-associated PAH, schistosomiasis associated PAH, PAH associated with portal hypertension, or pulmonary veno-occlusive disease (PVOD).
6. Recent history of left-sided heart disease and/or clinically significant cardiac disease within 48 weeks of Screening.
7. Left ventricular ejection fraction (LVEF) ≤ 50% within 24 weeks of Screening.
8. Hemodynamically significant valvular heart disease or uncontrolled symptomatic coronary disease.
9. History of atrial septostomy.
10. Uncontrolled atrial fibrillation or paroxysmal atrial fibrillation.
11. Untreated severe obstructive sleep apnea.
12. Hepatic dysfunction defined as Child-Pugh Class A or higher, or as evidenced by one of the following at Screening: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 x upper limit of normal (ULN) or total bilirubin ≥ 1.5 x ULN.
13. Severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or IP administration (eg, history of intracranial hemorrhage, recurrent syncope).
14. Any musculoskeletal disease, injury, or any other disease that limits evaluation of 6MWT.
15. Initiation of an exercise program for cardiopulmonary rehabilitation within 12 weeks prior to Screening or planned during the study.
16. Pregnant or nursing or intends to become pregnant during the duration of the study.
17. Body weight < 37 kg at Screening.
18. Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m^2 Hemoglobin (Hgb) concentration < 8.5 g/dL at Screening.
19. Evidence of active or latent Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C, or tuberculosis (TB) infection at Screening.
20. Prior/concurrent treatment with tyrosine kinase inhibitors or activin signaling inhibitors:

    1. Tyrosine kinase inhibitors, other than Janus kinase inhibitors approved for systemic autoimmune rheumatic diseases, within 12 weeks prior to Screening.
    2. Activin signaling inhibitors within 5 half-lives prior to Screening.
21. Requirement of IV inotropes (ie, levosimendan, dopamine, dobutamine, milrinone, norepinephrine) or IV diuretics for more than 24 hours within 4 weeks prior to Screening.
22. Subjects currently receiving oral anticoagulants (ie, warfarin/other vitamin K antagonists or direct-acting oral anticoagulants [DOACs]) if any of the following criteria are met:

    a. History within 24 weeks of Screening of: i. Syncope, or ii. Symptomatic bleeding in a critical area or organ iii. Intramuscular with compartment syndrome, or iv. Bleeding causing a fall in hemoglobin levels of 1.24 mmol/L (20 g/L or greater) or more, or v. Bleeding leading to a transfusion of 2 U or more of whole blood or red blood cells.

    b. History of central nervous system pathology.

    c. History of clinically significant (massive) hemoptysis.

    d. If on warfarin/other vitamin K antagonist, uncontrolled International normalized ratio (eg, INR > 3) as assessed.

    e. Platelet count < 150 x 10^9/L at Screening.

    f. Concomitant use of antiplatelet agents.

    g. CTD-APAH

    h. Concomitant use of sotatercept.
23. Prior participation in seralutinib studies and/or prior treatment with seralutinib.
24. Currently participating in or has participated in a study of an investigational agent or has used an investigational device for the treatment of PAH within 12 weeks or 5 half-lives of the investigational agent, whichever is longer, prior to Screening.
25. Current use of inhaled tobacco- or nicotine-containing products (including e-vapor products) and/or inhaled marijuana.
26. Current alcohol use disorder based on the opinion of the Investigator, and/or a positive test for drugs of abuse.
27. Subjects with a history of severe milk protein allergy or known intolerance to lactose.
28. QT interval corrected for heart rate using Fridericia's formula (QTcF) of > 500 msec.
29. Have any other condition or reason that, in the opinion of the Investigator or in the opinion of the Sponsor's Medical Monitor (MM) (or designee) in consultation with the Investigator, would prohibit the subject from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Change in distance achieved on the six-minute walk test (6MWT), six-minute walk distance (Δ6MWD) from baseline to Week 24 | Baseline to 24 weeks

SECONDARY OUTCOMES:
Time to first event of Clinical Worsening from first dose of Investigational Product (IP) through end of study | Baseline to 48 weeks
Proportion of subjects who achieve all of the following components of clinical improvement at Week 24, in the absence of clinical worsening: | Baseline to 24 weeks
  1. Improvement from baseline in World Health Organization (WHO) functional class (FC) or maintenance of WHO FC II
  2. Decrease from baseline in N-terminal pro b-type natriuretic peptide (NT-proBNP) of ≥ 30% or decrease and maintenance at < 300 ng/L
  3. Increase from baseline in 6MWD of ≥ 10% or ≥ 30 m
Change in NT-proBNP from baseline to Week 24 | Baseline to 24 weeks
Proportion of subjects with ≥ 1 point decrease from baseline in US Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) Lite 2 Risk Score at Week 24 | Baseline to 24 weeks
Proportion of subjects with each of the Clinical Worsening Outcomes: | Baseline to 52 weeks
  1. Death (all causes)
  2. Hospitalization for signs and symptoms of worsening PAH (≥ 24 hours)
  3. Worsening-related listing for or receipt of lung and/or heart/lung transplantation
  4. Atrial septostomy performed
  5. Worsening PAH requiring initiation of therapy with an additional approved background PAH disease-specific medication or the need to increase the dose of parenteral (IV or subcutaneous infusion) prostacyclin by 10% or more
  6. Disease progression, defined by both of the following events occurring at any time, even if they began at different times, as compared to their baseline values:
     1. Decrease in 6MWD of ≥ 15% on two consecutive tests, performed a minimum of 4 hours but no more than 1 week apart AND
     2. Worsened WHO FC
Proportion of subjects who improve from baseline in WHO FC or maintain WHO FC II | Baseline to 24 weeks
Change in PAH-SYMPACT™ from baseline to Week 24 | Baseline to 24 weeks
Change in Euro-QoL - 5 Dimensions - 5 Levels (EQ-5D-5L) from baseline to Week 24 | Baseline to 24 weeks
Incidence of treatment-emergent adverse events (TEAEs), serious TEAEs (SAEs), and treatment-emergent adverse events of special interest (AESIs) | Baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aranda, MD, Study Director — Gossamer Bio Inc.
Locations (166):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valley Advanced Lung Diseases Institute, Fresno, California
  - Keck Medical Center of USC, Los Angeles, California
  - Dept of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - UC Davis Health, Sacramento, California
  - Stanford Healthcare, Stanford, California
  - Winchester Center for Lung Disease, New Haven, Connecticut
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Piedmont Physicians Pulmonary & Sleep Medicine of Buckhead, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northside Hospital Laboratory - Atlanta, Atlanta, Georgia
  - UI Health Hospital, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Hospital, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center - Duke South, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - INTEGRIS Cardiovascular Physicians, LLC, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple Heart and Vascular Institute (Outpatient Clinic), Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina - Nexus Research Center, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Outpatient Center, Houston, Texas
  - Baylor Scott & White Medical Center - The Heart Hospital, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Advocate Aurora Health-Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (8):
  - Cardiologia Palermo, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - Hospital Privado Centro Medico de Cordóba S.A., Córdoba
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Sanatorio Parque S.A., Rosario
  - Hospital Provincial Dr. José María Cullen, Santa Fe
- Australia (4):
  - St Vincent's Hospital, Melbourne, Victoria
  - Wesley Research Institute, Auchenflower
  - Royal Hobart Hospital, Hobart
  - Nepean Hospital, Kingswood
- Austria (2):
  - Religious Hospital Linz GmbH, Linz
  - AKH-Vienna Medical Univesity of Vienna Internal Medicine II-Cardiology, Vienna
- Belgium (2):
  - Hôpital Erasme, Anderlecht
  - University Hospitals of Leuven (Campus Gasthuisberg), Leuven
- Brazil (6):
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Complexo de Prevencao, Diagnostico, Terapia e Reabilitacao Respiratoria - Hospital Dia do Pulmao, Blumenau
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educaçao e Assistência Hospital São Lucas da PUCRS, Porto Alegre
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Núcleo de Gestão de Pesquisa/Hospital São Paulo - SPDM/UNIFESP, São Paulo
- Canada (4):
  - London Health Science Centre - Victoria Hospital, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Peter Lougheed Center, Calgary
  - University Health Network, Toronto
- Chile (2):
  - Enroll SpA, Santiago, Santiago Metropolitan
  - Centro de Investigacion Clinica UC-CICUC, Santiago
- Colombia (2):
  - Fundación Abood Shaio, Bogotá
  - Fundación Neumologica Colombiana, Bogotá
- Czechia (2):
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Všeobecná fakultní nemocnice v Praze Il. interní klinika kardiologie a angiologie VFN a 1.LF UK Centrum pro plicní hypertenzi, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Department of Cardiology, Aarhus
  - Rigshospitalet, Department of Cardiology, Copenhagen
- France (7):
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Institut Coeur Poumon, Lille
  - CHU de Montpellier, Montpellier
  - Hôpital Pasteur, Nice
  - CHU de Poitiers, Poitiers
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire - Hôpital d´Adultes de Brabois, Vandœuvre-lès-Nancy
- Germany (10):
  - DRK Kliniken Berlin Westend, Berlin
  - Zentrum fur Pulmona le Hypertonie, Klini k Ill fur lnnere Medizin (Kardiologie, Pneumologie, lnternlstische lntensiv medizin), Herzzentrum der Universitat zu Koln, Cologne
  - Universitatsklinikum Dresden, Medizinische Klinik / Pneumologisches Studiensekretariat, Dresden
  - Universitatsklinikum Giessen und Marburg GmbH Zentrum fur Innere Medizin, Med. Klinik und Poliklinik II Studienambulanz fur Pulmonale Hypertonie, Giessen
  - Universitätsklinikum Greifswald Klinik und Poliklinik für Innere Medizin B, Greifswald
  - Universitätsklinikum Halle (Saale) / Martin-Luther-Universität Halle- Wittenberg, Universitätsklinik und Poliklinik für Innere Medizin I, Halle
  - Thoraxklinik Heidelberg gGmbH am Universitätsklinikum Heidelberg Zentrum für pulmonale Hypertonie, Heidelberg
  - Krankenhaus Neuwittelsbach, Munich
  - Klinikum der LMU Medizinische Klinik und Poliklinik V, München
  - Klinikum Wurzburg Mitte gGmbH Medizinische Klinik mit Schwerpunkt Pneumologie und Beatmungsmedizin, Würzburg
- Greece (4):
  - "Evangelismos" General Hospital, 1st Department of Clinical Care & Pulmonary Hypertension Clinic, Athens
  - ATTIKON University Hospital, 2nd Critical Care Department, Athens
  - Onassis Cardiac Surgery Center, Kallithea
  - AHEPA University General Hospital of Thessaloniki, 1st Cardiology Clinic, Thessaloniki
- Mater Misericordiae University Hospital, Respiratory Department, Dublin, Ireland
- Israel (5):
  - Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - IRCCS Azienda Ospedaliero Universitaria Di Bologna Policlinico 5 Orsola Malpighi - U.O.C. Cardiologia, Bologna
  - Azienda Ospedaliera Dei Colli - Ospedale Monaldi Centro per la Diagnosi e Terapia dell'Ipertensione Polmonare, Napoli
  - Fondazione IRCCS Policlinico San Matteo - U.O. di Cardiologia, Pavia
  - Azienda Ospealiero Universitaria Policlinico Umberto I - Dipartamento di Scienze Cliniche Internistiche Anestesiologiche e Cardiovascolari - VIII Padglione, Rome
  - Azienda Sanitaria Universitaria Giuliano Isontina /ASUGI - Ospedale di Cattinara - Cardiovascular Department Coronary Intensive Care Unit, Trieste
- Japan (8):
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Kurume
  - Nagoya University Hospital, Nagoya
  - NHO Okayama Medical Center, Okayama
  - Keio University Hospital, Shinjuku-Ku
  - National Cerebral and Cardiovascular Center, Suita
  - Kyorin University Hospital, Tokyo
  - University of Tokyo Hospital, Tokyo
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Mexico (3):
  - Instituto nacional de Cardiologia Ignacio Chavez, Mexico City
  - Hospital Universitario Dr. José Eleuterio González Centro de Prevención y Rehabilitación de Enfermedades Pulmonares Crónicas, Monterrey
  - Unidad de Investigacion Clinica en Medicina, S.C., Monterrey
- Netherlands (2):
  - Amsterdam UMC, location VUmc, Amsterdam
  - Erasmus MC, Rotterdam
- Poland (2):
  - Krakowski Szpital Specjalistyczny Im. Św. Jana Pawła II Oddział Kliniczny Chorób Serca i Naczyń z Pododdziałem Intensywnego Nadzoru Kardiologicznego, Krakow
  - Europejskie Centrum Zdrowia Otwock Sp. z o.o. Szpital irn. Fryderyka Chopina Oddzial Kardiologiczny, Otwock
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Centro Hospitalar Universitário Lisboa Norte, EPE - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar Universitário de Santo António, Porto
- Romania (4):
  - Emergency Institute of Cardiovascular Diseases "Prof. Dr. C.C. Iliescu" Bucharest, Cardiology 2, Bucharest
  - "Niculae Stanciolu" Emergency Heart Institute for Cardivascular Diseases, Cluj-Napoca
  - Mediprax Centrum S.R.L, Cluj-Napoca
  - Targu-Mures Emergency Clinical County Hospital, Internal Medicine II, Târgu Mureş
- Saudi Arabia (2):
  - King Fahad Medical City, Riyadh
  - King Faisal Specialist Hospital and Research Center, Riyadh
- Serbia (2):
  - Institute for Cardiovascular Diseases "Dedinje" Clinic for Cardiology, Belgrade
  - University Clinical Centre of Serbia, Cardiology Clinic, Belgrade
- Singapore (2):
  - National Heart Centre Singapore, Singapore
  - National University Heart Centre Singapore, Singapore
- South Korea (5):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System Seoul, Seoul
  - The Catholic University of Korea, Seoul St. Mary´s Hospital, Seoul
- Spain (8):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Puerta De Hierro Majadahonda, Majadahonda
  - Hospital Costa del Sol, Marbella
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Toledo, Toledo
- United Kingdom (7):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Golden Jubilee National Hospital, Agamemnon Street, Clydebank
  - Hammersmith Hospital, London
  - Royal Brompton Hospital, Pulmonary Hypertension Service, Sydney Street, London
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle
  - Sheffield Clinical Research Facility, Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sitbon O, Sahay S, Escribano Subias P, Zolty RL, Kingrey JF, Ryan JJ, Sobol I, Sood N, Benza RL, Channick RN, Chin KM, Frantz RP, Ghofrani HA, Hemnes AR, McLaughlin VV, Vachiery JL, Zamanian RT, Ter Veer A, Roscigno RF, Mottola D, Parsley E, Aranda R, Zisman LS, Howard LS; TORREY Study Investigators. Seralutinib for the Treatment of Pulmonary Arterial Hypertension in Adults: TORREY Open-Label Extension Study. Adv Ther. 2025 Oct;42(10):5104-5123. doi: 10.1007/s12325-025-03297-2. Epub 2025 Aug 11. PMID 40788460